CLINICAL TRIAL: NCT03522051
Title: Assessment of Pulpotomy Procedure Using NeoMTA Plus in Permanent Teeth With Carious Exposure
Acronym: PULPOTOMY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JUST14-4-2018
Record Dates: First submitted 2018-04-19; First posted 2018-05-11 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Pulpotomy
Keywords: teeth; pulpitis; deep caries; pulpotomy; Mineral Trioxide Aggregate (MTA)
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Intervention Model Description: Patients with symptomatic deep caries in a permanent molar tooth will receive pulpotomy treatment and placement of a calcium silicate based material (Neo MTA plus) over the pulp and followed by restoration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with carious teeth (Experimental): female or male patients with permanent teeth and deep caries will receive pulpotomy treatment and dressing with calcium silicate based material (Neo MTA plus material) followed by restoration.
  Interventions: Other: calcium silicate based material,

INTERVENTIONS:
Other: calcium silicate based material, — Its a dental pulp capping material which is biocompatable and induces hard tissue barrier formation
  Other Names: Neo MTA plus, Avalon Biomed

SUMMARY:
Many deep carious teeth are treated unnecessarily by root canal therapy, while with using current techniques and advances in compatible dental materials in addition to better understanding of biological response of the dental pulp, many can be treated conservatively via vital pulp therapy procedures.

DETAILED DESCRIPTION:
Vital pulp therapy is recommended for teeth diagnosed with reversible pulpitis or partially inflamed pulps in which the remaining healthy tissue can be conserved and protected by a biologically active material to generate a hard tissue barrier that seals and protects the pulp from future microbial insult.

The aim of this in vivo study is to clinically and radiographically assess the outcome of full pulpotomy using a calcium silicate based material (NeoMTA Plus) in permanent teeth with carious exposure.

Ethics approval was obtained from the institutional ethics and research committee, and the patients were informed about details of the treatment and the possible complications. An informed consent was obtained. 120 patients meeting the inclusion criteria will be selected for this study and they will be subsequently followed up clinically and radiographically after 3 months, 6 months, 1 year and yearly afterward for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Permanent teeth with mature or immature apices
* Have no significant medical problems
* The tooth should give positive response to cold test and electric pulp test (EPT)
* Probing pocket depth and mobility within normal limits
* No Signs of pulp necrosis including sinus tract or swelling
* Radiographically ; caries either exposing the pulps or reaching more than 2\3 the distance from the dentino-enamel junction (DEJ) to the pulp
* The tooth can be restored via direct restoration

Exclusion Criteria:

* Medically compromised patients
* Negative response to cold test
* Mobility
* Sinus tract
* Swelling
* Non restorable teeth or badly broken teeth

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Change in pain symptoms | 2-3 days after the treatment, 3 months, 6 months and 12 months and afterwards up to 5 years.
  The patient is anticipated to report reduction in the pain score after receiving the treatment within 2-3 days and the tooth should continue to be asymptomatic at follow up appointments. The patient will be asked to score the pain level on visual analogue scale using a score from 0-10. The zero is no pain while 10 is the maximum level.

SECONDARY OUTCOMES:
Periapical normalcy at follow up radiographs . | 6months , 1 year, 2, 3,4,5 years
  Pr-existing pathology should heal within 6 months- 1 year and normalcy should be maintained after ward up to 5 years.
  no emerging pathosis should be evident in the roots or surrounding bone.
The tooth and restoration should be present in the mouth | 3, 6 months, 1 year, 2, 3,4,5 years
  The tooth should be in the mouth and in function (not extracted) with an intact restoration at the follow up times

CONTACTS AND LOCATIONS:
Overall Officials: Nessrin A Taha, PhD, Study Director — Jordan University of Science and Technology
Locations (1):
- Jordan University of science and technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
Baseline demographic data and follow-up results may be shared after manuscript acceptance by international journals

REFERENCES:
- [Background] Taha NA, Abdelkhader SZ. Outcome of full pulpotomy using Biodentine in adult patients with symptoms indicative of irreversible pulpitis. Int Endod J. 2018 Aug;51(8):819-828. doi: 10.1111/iej.12903. Epub 2018 Feb 27. PMID 29397003
- [Background] Taha NA, Khazali MA. Partial Pulpotomy in Mature Permanent Teeth with Clinical Signs Indicative of Irreversible Pulpitis: A Randomized Clinical Trial. J Endod. 2017 Sep;43(9):1417-1421. doi: 10.1016/j.joen.2017.03.033. Epub 2017 Jun 30. PMID 28673494
- [Background] Taha NA, Ahmad MB, Ghanim A. Assessment of Mineral Trioxide Aggregate pulpotomy in mature permanent teeth with carious exposures. Int Endod J. 2017 Feb;50(2):117-125. doi: 10.1111/iej.12605. Epub 2016 Jan 30. PMID 26715408

DOCUMENTS (1):
  • Study Protocol (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT03522051/Prot_000.pdf